CLINICAL TRIAL: NCT05504616
Title: Physical Activity in Axial Spondyloarthritis: Development and Implementation of an Evidence-Based Health Technology Approach to Improve Adherence to Recommended Guidelines
Brief Title: Health Technology to Improve Exercise in axSpA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Initiative for Outcomes in Rheumatology Care (Other)
Responsible Party: Principal Investigator, Laura Passalent, Physiotherapist Practitioner, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-5919
Record Dates: First submitted 2022-07-29; First posted 2022-08-17 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Intervention Model Description: Repeated measures randomized control pre-test/post-test design comparing an intervention group with a control group (usual care).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants randomized to the intervention group will receive an initial electronic communication (i.e. email) that includes:
  * Link to physical activity education. This will be an educational module based on Phase 1 results and evidence-based literature regarding the benefits of physical activity in the general population and specific to axSpA.
  * One week after receiving the physical activity educational module, participants will receive access to the ADAS application and an .ics file for each 3-week cycle of electronic calendar reminders to engage in physical activity.
  Interventions: Other: Health technology-based intervention strategy
- Control Group (No Intervention): Participants randomized to the control group will receive usual care, which includes standard rheumatology care and access to educational materials on the importance of exercise and physical activity available through the TWH Spondylitis Program and through the public domain. They will receive a link to the physical activity educational module at baseline. They also have access to the program physiotherapist for a single one-hour individualized exercise consultation as requested by either the patient or the treating rheumatologist.

INTERVENTIONS:
Other: Health technology-based intervention strategy — Patient-centered, technology-based intervention strategy aimed at increasing physical activity in patients with axSpA
  Arms: Intervention Group

SUMMARY:
Despite the known benefits of physical activity, the majority of Canadians fail to meet recommended guidelines. Patients with axial spondyloarthritis (axSpA) also fail to meet recommended guidelines. Exercise, a critical component of physical activity, is considered the cornerstone of axSpA management. Simple health technologies such as mobile phone messaging and email can be useful tools to increase engagement in regular physical activity among the general public and patients with chronic disease. As such, the aim of this research project is to develop and test a patient-centered strategy that provides education on the importance of physical activity and utilizes existing health technologies (such as smart phone applications) to encourage regular participation in physical activity. The results of this study are expected to demonstrate that patients with axSpA will increase their daily engagement in physical activity, and therefore improve symptoms, function and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18 and older) with a diagnosis of axSpA based on ASAS criteria
* Have access to email and a smart phone device (Android or iOS operating systems)
* Enrolled in the SPARCC Research Program
* Passes pre-participation health screen

Exclusion Criteria:

* Non-English speaking
* Not enrolled in the SPARCC Research Program
* Comorbidities or physical impairments that may preclude physical activity (e.g., symptomatic cardiovascular disease; wheelchair bound etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in levels of physical activity as measured by the International Physical Activity Questionnaire-Short Form questionnaire (IPAQ-SF) | Assessed electronically by an e-survey platform at baseline, 3, 6, 9 and 12 weeks in the intervention and control groups.
  The IPAQ-SF is a self-report questionnaire designed to estimate total physical activity in MET-min/week by assessing the types of intensity of physical activity and sitting time that people do as part of their daily lives.
Changes in exercise behaviour as measured by an adapted Stanford Exercise Behaviours Questionnaire | Assessed electronically by an e-survey platform at baseline, 3, 6, 9 and 12 weeks in the intervention and control groups.
  2-item questionnaire measuring total time (minutes) spent on stretching and strengthening exercises each week.
Change in levels of physical activity as measured by Accelerometry | Assessed at baseline and at 12 weeks.
  Participants wear an accelerometer for 7 consecutive days at baseline and again at 12 weeks. The participant will mail back the activity monitor using a pre-paid envelope following each seven-day period.
Change in perceived benefits and barriers to exercise as a result of the technology-based intervention strategy as measured by the Exercise Benefits/Barriers Scale (EBBS) | Assessed at baseline and at 12 weeks.
  The EBBS measures perceptions regarding the benefits of, and barriers to, exercise.
Change in functioning and health as a result of the technology-based intervention strategy as measured by the ASAS Health Index | Assessed at baseline and at 12 weeks.
  The self-report questionnaire measures functioning and health across 17 aspects of health and 9 environmental factors in patients with spondyloarthritis. The items measure the concept of 'functioning, disability and health'

SECONDARY OUTCOMES:
Change in disease activity over the course of 12 weeks as measured by the Bath Ankylosing Spondylitis Disease Activity Index (BASDI) questionnaire | From baseline, assessed up to 12 weeks.
  Disease activity, including pain, fatigue and stiffness as measured by the BASDAI questionnaire (a 0 - 10 visual analog scale) weekly.
Change in function over the course of 12 weeks as measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) questionnaire | From baseline, assessed up to 12 weeks.
  Function as measured by the BASFI questionnaire (0 - 10 visual analog scale) weekly.
Number of accepted invites over the course of 12 weeks | From baseline, assessed up to 12 weeks.
  Acceptance of planned exercise, as measured by uptake of health technology-based intervention strategy
Frequency of physical activity sessions as a result of the technology-based intervention strategy over the course of 12 weeks | From baseline, assessed up to 12 weeks.
  Acceptance of planned exercise, as measured by uptake of health technology-based intervention strategy
Duration of physical activity sessions as a result of the technology-based intervention strategy over the course of 12 weeks | From baseline, assessed up to 12 weeks.
  Acceptance of planned exercise, as measured by uptake of health technology-based intervention strategy
Acceptance of health technology-based intervention strategy, as measured by the Mobile Application Rating Scale | Assessed at 12 weeks.
  Acceptance of intervention, as measured by the Mobile Application Rating Scale. MARS is a 5-point scale from 1-inadequate or strongly disagree to 5-excellent or strongly agree that accesses app quality, app subjective quality, and perceived impact of the app on user's knowledge, intentions to change as well as the likelihood of actual change in the target health behaviour. Higher scores indicate greater quality and acceptance of the intervention.
Number of enrolled participants who complete the study | Assessed at 12 weeks.
  Adherence, as measured by the rate of study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Passalent, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network - Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. World Health Organization. Fact Sheet Updated February 2018. Available at: http://www.who.int/mediacentre/factsheets/fs385/en/ Accessed on March 26, 2018
- [Background] Canadian Society for Exercise Physiology. Canadian physical activity guidelines. 2011. Available at http://www.csep.ca/CMFiles/Guidelines/CanadianPhysicalActivityGuidelinesStatements_E%203.pdf. Accessed on March 29, 2018
- [Background] World Health Organization. Physical activity. Available at: http://www.who.int/topics/physical_activity/en/ Accessed on March 29, 2018
- [Background] Sieper J, Rudwaleit M, Baraliakos X, Brandt J, Braun J, Burgos-Vargas R, Dougados M, Hermann KG, Landewe R, Maksymowych W, van der Heijde D. The Assessment of SpondyloArthritis international Society (ASAS) handbook: a guide to assess spondyloarthritis. Ann Rheum Dis. 2009 Jun;68 Suppl 2:ii1-44. doi: 10.1136/ard.2008.104018. PMID 19433414
- [Background] Dagfinrud H, Kvien TK, Hagen KB. Physiotherapy interventions for ankylosing spondylitis. Cochrane Database Syst Rev. 2008 Jan 23;2008(1):CD002822. doi: 10.1002/14651858.CD002822.pub3. PMID 18254008
- [Background] van der Heijde D, Ramiro S, Landewe R, Baraliakos X, Van den Bosch F, Sepriano A, Regel A, Ciurea A, Dagfinrud H, Dougados M, van Gaalen F, Geher P, van der Horst-Bruinsma I, Inman RD, Jongkees M, Kiltz U, Kvien TK, Machado PM, Marzo-Ortega H, Molto A, Navarro-Compan V, Ozgocmen S, Pimentel-Santos FM, Reveille J, Rudwaleit M, Sieper J, Sampaio-Barros P, Wiek D, Braun J. 2016 update of the ASAS-EULAR management recommendations for axial spondyloarthritis. Ann Rheum Dis. 2017 Jun;76(6):978-991. doi: 10.1136/annrheumdis-2016-210770. Epub 2017 Jan 13. PMID 28087505
- [Background] Ward MM, Deodhar A, Akl EA, Lui A, Ermann J, Gensler LS, Smith JA, Borenstein D, Hiratzka J, Weiss PF, Inman RD, Majithia V, Haroon N, Maksymowych WP, Joyce J, Clark BM, Colbert RA, Figgie MP, Hallegua DS, Prete PE, Rosenbaum JT, Stebulis JA, van den Bosch F, Yu DT, Miller AS, Reveille JD, Caplan L. American College of Rheumatology/Spondylitis Association of America/Spondyloarthritis Research and Treatment Network 2015 Recommendations for the Treatment of Ankylosing Spondylitis and Nonradiographic Axial Spondyloarthritis. Arthritis Rheumatol. 2016 Feb;68(2):282-98. doi: 10.1002/art.39298. Epub 2015 Sep 24. PMID 26401991
- [Background] Rausch Osthoff AK, Niedermann K, Braun J, Adams J, Brodin N, Dagfinrud H, Duruoz T, Esbensen BA, Gunther KP, Hurkmans E, Juhl CB, Kennedy N, Kiltz U, Knittle K, Nurmohamed M, Pais S, Severijns G, Swinnen TW, Pitsillidou IA, Warburton L, Yankov Z, Vliet Vlieland TPM. 2018 EULAR recommendations for physical activity in people with inflammatory arthritis and osteoarthritis. Ann Rheum Dis. 2018 Sep;77(9):1251-1260. doi: 10.1136/annrheumdis-2018-213585. Epub 2018 Jul 11. PMID 29997112
- [Background] Haroon NN, Paterson JM, Li P, Inman RD, Haroon N. Patients With Ankylosing Spondylitis Have Increased Cardiovascular and Cerebrovascular Mortality: A Population-Based Study. Ann Intern Med. 2015 Sep 15;163(6):409-16. doi: 10.7326/M14-2470. PMID 26258401
- [Background] Klingberg E, Lorentzon M, Mellstrom D, Geijer M, Gothlin J, Hilme E, Hedberg M, Carlsten H, Forsblad-d'Elia H. Osteoporosis in ankylosing spondylitis - prevalence, risk factors and methods of assessment. Arthritis Res Ther. 2012 May 8;14(3):R108. doi: 10.1186/ar3833. PMID 22569245
- [Background] Feldtkeller E, Vosse D, Geusens P, van der Linden S. Prevalence and annual incidence of vertebral fractures in patients with ankylosing spondylitis. Rheumatol Int. 2006 Jan;26(3):234-9. doi: 10.1007/s00296-004-0556-8. Epub 2005 Mar 11. PMID 15761730
- [Background] Dursun N, Sarkaya S, Ozdolap S, Dursun E, Zateri C, Altan L, Birtane M, Akgun K, Revzani A, Aktas I, Tastekin N, Celiker R. Risk of falls in patients with ankylosing spondylitis. J Clin Rheumatol. 2015 Mar;21(2):76-80. doi: 10.1097/RHU.0000000000000216. PMID 25710858
- [Background] Passalent LA, Soever LJ, O'Shea FD, Inman RD. Exercise in ankylosing spondylitis: discrepancies between recommendations and reality. J Rheumatol. 2010 Apr;37(4):835-41. doi: 10.3899/jrheum.090655. Epub 2010 Mar 1. PMID 20194443
- [Background] Arturi P, Schneeberger EE, Sommerfleck F, Buschiazzo E, Ledesma C, Maldonado Cocco JA, Citera G. Adherence to treatment in patients with ankylosing spondylitis. Clin Rheumatol. 2013 Jul;32(7):1007-15. doi: 10.1007/s10067-013-2221-7. Epub 2013 Mar 21. PMID 23515597
- [Background] Swinnen TW, Scheers T, Lefevre J, Dankaerts W, Westhovens R, de Vlam K. Physical activity assessment in patients with axial spondyloarthritis compared to healthy controls: a technology-based approach. PLoS One. 2014 Feb 28;9(2):e85309. doi: 10.1371/journal.pone.0085309. eCollection 2014. PMID 24586239
- [Background] O'Dwyer T, O'Shea F, Wilson F. Physical activity in spondyloarthritis: a systematic review. Rheumatol Int. 2015 Mar;35(3):393-404. doi: 10.1007/s00296-014-3141-9. Epub 2014 Oct 10. PMID 25300728
- [Background] O'Dwyer T, McGowan E, O'Shea F, Wilson F. Physical Activity and Exercise: Perspectives of Adults With Ankylosing Spondylitis. J Phys Act Health. 2016 May;13(5):504-13. doi: 10.1123/jpah.2015-0435. Epub 2015 Oct 28. PMID 26529384
- [Background] Jahangiry L, Farhangi MA, Shab-Bidar S, Rezaei F, Pashaei T. Web-based physical activity interventions: a systematic review and meta-analysis of randomized controlled trials. Public Health. 2017 Nov;152:36-46. doi: 10.1016/j.puhe.2017.06.005. Epub 2017 Jul 20. PMID 28734170
- [Background] Marcolino MS, Oliveira JAQ, D'Agostino M, Ribeiro AL, Alkmim MBM, Novillo-Ortiz D. The Impact of mHealth Interventions: Systematic Review of Systematic Reviews. JMIR Mhealth Uhealth. 2018 Jan 17;6(1):e23. doi: 10.2196/mhealth.8873. PMID 29343463
- [Background] Mayer JE, Fontelo P. Meta-analysis on the effect of text message reminders for HIV-related compliance. AIDS Care. 2017 Apr;29(4):409-417. doi: 10.1080/09540121.2016.1214674. Epub 2016 Aug 1. PMID 27477580
- [Background] Foster C, Richards J, Thorogood M, Hillsdon M. Remote and web 2.0 interventions for promoting physical activity. Cochrane Database Syst Rev. 2013 Sep 30;9(9):CD010395. doi: 10.1002/14651858.CD010395.pub2. PMID 24085594
- [Background] Tyrrell JS, Redshaw CH. Physical Activity in Ankylosing Spondylitis: evaluation and analysis of an eHealth tool. J Innov Health Inform. 2016 Jul 4;23(2):169. doi: 10.14236/jhi.v23i2.169. PMID 27869581
- [Background] Griffiths AJ, White CM, Thain PK, Bearne LM. The effect of interactive digital interventions on physical activity in people with inflammatory arthritis: a systematic review. Rheumatol Int. 2018 Sep;38(9):1623-1634. doi: 10.1007/s00296-018-4010-8. Epub 2018 Mar 19. PMID 29556750
- [Background] Kang R, Passalent L, Morton R, Hawke C, Blair J, Lake A, et al. The European league against rheumatism (EULAR) 2013. Utilization of an informational needs assessment to develop an education program for patients with ankylosing spondylitis and related axial spondyloarthritis
- [Background] Haglund E, Bremander A, Bergman S, Larsson I. Educational needs in patients with spondyloarthritis in Sweden - a mixed-methods study. BMC Musculoskelet Disord. 2017 Aug 2;18(1):335. doi: 10.1186/s12891-017-1689-8. PMID 28768510
- [Background] Rudwaleit M, van der Heijde D, Landewe R, Listing J, Akkoc N, Brandt J, Braun J, Chou CT, Collantes-Estevez E, Dougados M, Huang F, Gu J, Khan MA, Kirazli Y, Maksymowych WP, Mielants H, Sorensen IJ, Ozgocmen S, Roussou E, Valle-Onate R, Weber U, Wei J, Sieper J. The development of Assessment of SpondyloArthritis international Society classification criteria for axial spondyloarthritis (part II): validation and final selection. Ann Rheum Dis. 2009 Jun;68(6):777-83. doi: 10.1136/ard.2009.108233. Epub 2009 Mar 17. PMID 19297344
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qualitative Research In Psychology 2008;3(2):77-101
- [Background] Fanning J, Mullen SP, McAuley E. Increasing physical activity with mobile devices: a meta-analysis. J Med Internet Res. 2012 Nov 21;14(6):e161. doi: 10.2196/jmir.2171. PMID 23171838
- [Background] Orr JA, King RJ. Mobile phone SMS messages can enhance healthy behaviour: a meta-analysis of randomised controlled trials. Health Psychol Rev. 2015;9(4):397-416. doi: 10.1080/17437199.2015.1022847. Epub 2015 May 28. PMID 25739668
- [Background] Stock MS, Mota JA, DeFranco RN, Grue KA, Jacobo AU, Chung E, Moon JR, DeFreitas JM, Beck TW. The time course of short-term hypertrophy in the absence of eccentric muscle damage. Eur J Appl Physiol. 2017 May;117(5):989-1004. doi: 10.1007/s00421-017-3587-z. Epub 2017 Mar 20. PMID 28321637
- [Background] Miller MG, Herniman JJ, Ricard MD, Cheatham CC, Michael TJ. The effects of a 6-week plyometric training program on agility. J Sports Sci Med. 2006 Sep 1;5(3):459-65. eCollection 2006. PMID 24353464
- [Background] Seynnes OR, de Boer M, Narici MV. Early skeletal muscle hypertrophy and architectural changes in response to high-intensity resistance training. J Appl Physiol (1985). 2007 Jan;102(1):368-73. doi: 10.1152/japplphysiol.00789.2006. Epub 2006 Oct 19. PMID 17053104
- [Background] American College of Sports Medicine Exercise pre-participation health screening recommendations. 2015 Available at: http://www.acsm.org/docs/default-source/publications/acsm-101-prescreeninginfographiccolorlegal-2015-12-15-v02.pdf?sfvrsn=2 . Accessed on March 28, 2018
- [Background] Passalent L, Kang R, Lawson D, Hawke C, Omar A, Thavaneswaran A, Haroon N, Inman RD. Impact of e-learning on knowledge, self-efficacy and exercise behaviours in patients with axial spondyloarthritis: results from a longitudinal randomized control trial [abstract]. Arthritis Rheumatol. 2016;68 (suppl 10)
- [Background] Lawson D, Passalent L, Kang R, Hawke C, Omar A, Thavaneswaran A, Haroon N, Inman RD. Impact of e-learning on perceived social role participation of patients with axial spondyloarthritis: results from a longitudinal randomized control train [abstract]. Arthritis Rheumatol. 2016;68 (suppl 10)
- [Background] Kim J, Shin W. How to do random allocation (randomization). Clin Orthop Surg. 2014 Mar;6(1):103-9. doi: 10.4055/cios.2014.6.1.103. Epub 2014 Feb 14. PMID 24605197
- [Background] Wendel-Vos GC, Schuit AJ, Saris WH, Kromhout D. Reproducibility and relative validity of the short questionnaire to assess health-enhancing physical activity. J Clin Epidemiol. 2003 Dec;56(12):1163-9. doi: 10.1016/s0895-4356(03)00220-8. PMID 14680666
- [Background] Arends S, Hofman M, Kamsma YP, van der Veer E, Houtman PM, Kallenberg CG, Spoorenberg A, Brouwer E. Daily physical activity in ankylosing spondylitis: validity and reliability of the IPAQ and SQUASH and the relation with clinical assessments. Arthritis Res Ther. 2013 Aug 23;15(4):R99. doi: 10.1186/ar4279. PMID 23971767
- [Background] Lorig K, Stewart A, Ritter P, Gonzalez V, Laurent D, Lynch J. Outcome measures for health education and other health care interventions. Thousand Oaks, CA; Sage Publications, 1996, pp.25,37-38
- [Background] Sechrist KR, Walker SN, Pender NJ. Development and psychometric evaluation of the exercise benefits/barriers scale. Res Nurs Health. 1987 Dec;10(6):357-65. doi: 10.1002/nur.4770100603. PMID 3423307
- [Background] Neuberger GB, Kasal S, Smith KV, Hassanein R, DeViney S. Determinants of exercise and aerobic fitness in outpatients with arthritis. Nurs Res. 1994 Jan-Feb;43(1):11-7. PMID 8295833
- [Background] O'Dwyer T, Rafferty T, O'Shea F, Gissane C, Wilson F. Physical activity guidelines: is the message getting through to adults with rheumatic conditions? Rheumatology (Oxford). 2014 Oct;53(10):1812-7. doi: 10.1093/rheumatology/keu177. Epub 2014 May 14. PMID 24829221
- [Background] Fabre S, Molto A, Dadoun S, Rein C, Hudry C, Kreis S, Fautrel B, Pertuiset E, Gossec L. Physical activity in patients with axial spondyloarthritis: a cross-sectional study of 203 patients. Rheumatol Int. 2016 Dec;36(12):1711-1718. doi: 10.1007/s00296-016-3565-5. Epub 2016 Sep 24. PMID 27665288
- [Background] Oosterom N, Gant CM, Ruiterkamp N, van Beijnum BF, Hermens H, Bakker SJL, Navis G, Vollenbroek-Hutten MMR, Laverman GD. Physical Activity in Patients With Type 2 Diabetes: The Case for Objective Measurement in Routine Clinical Care. Diabetes Care. 2018 Apr;41(4):e50-e51. doi: 10.2337/dc17-2041. Epub 2018 Feb 6. No abstract available. PMID 29432126
- [Background] Trost SG, McIver KL, Pate RR. Conducting accelerometer-based activity assessments in field-based research. Med Sci Sports Exerc. 2005 Nov;37(11 Suppl):S531-43. doi: 10.1249/01.mss.0000185657.86065.98. PMID 16294116
- [Background] van der Heijde D, Calin A, Dougados M, Khan MA, van der Linden S, Bellamy N. Selection of instruments in the core set for DC-ART, SMARD, physical therapy, and clinical record keeping in ankylosing spondylitis. Progress report of the ASAS Working Group. Assessments in Ankylosing Spondylitis. J Rheumatol. 1999 Apr;26(4):951-4. PMID 10229426
- [Background] Garrett S, Jenkinson T, Kennedy LG, Whitelock H, Gaisford P, Calin A. A new approach to defining disease status in ankylosing spondylitis: the Bath Ankylosing Spondylitis Disease Activity Index. J Rheumatol. 1994 Dec;21(12):2286-91. PMID 7699630
- [Background] Calin A, Garrett S, Whitelock H, Kennedy LG, O'Hea J, Mallorie P, Jenkinson T. A new approach to defining functional ability in ankylosing spondylitis: the development of the Bath Ankylosing Spondylitis Functional Index. J Rheumatol. 1994 Dec;21(12):2281-5. PMID 7699629
- [Background] Doward LC, Spoorenberg A, Cook SA, Whalley D, Helliwell PS, Kay LJ, McKenna SP, Tennant A, van der Heijde D, Chamberlain MA. Development of the ASQoL: a quality of life instrument specific to ankylosing spondylitis. Ann Rheum Dis. 2003 Jan;62(1):20-6. doi: 10.1136/ard.62.1.20. PMID 12480664
- [Background] Hillsdon M, Foster C, Thorogood M. Interventions for promoting physical activity. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD003180. doi: 10.1002/14651858.CD003180.pub2. PMID 15674903
- [Background] O'Dwyer T, O'Shea F, Wilson F. Decreased physical activity and cardiorespiratory fitness in adults with ankylosing spondylitis: a cross-sectional controlled study. Rheumatol Int. 2015 Nov;35(11):1863-72. doi: 10.1007/s00296-015-3339-5. Epub 2015 Aug 9. PMID 26254884
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Zelenko O, Tjondronegoro D, Mani M. Mobile app rating scale: a new tool for assessing the quality of health mobile apps. JMIR Mhealth Uhealth. 2015 Mar 11;3(1):e27. doi: 10.2196/mhealth.3422. PMID 25760773